CLINICAL TRIAL: NCT05333744
Title: The Combination of Prednisone and Recombinant Human Thrombopoietin vs Prednisone Monotherapy for Treatment in Immune Thrombocytopenia in Pregnancy
Brief Title: The Combination of Prednisone and Recombinant Human Thrombopoietin for Treatment of Immune Thrombocytopenia in Pregnancy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-PKU2204
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone; Thrombopoietin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone plus rhTPO (Experimental): Prednisone 20mg per day, 2 weeks and rhTPO 300U/kg per day, 2 weeks
  Interventions: Drug: Prednisone; Drug: Recombinant Human TPO
- Prednisone (Active Comparator): Prednisone 20mg per day, 2 weeks
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone po, 20mg per day for 2 weeks, if response (Plt 30-100×100^g/L),gradually taper to the maintenance dose（5-10mg per day）until 6 weeks after delivery; if not response, gradually taper to withdrawal.
Drug: Recombinant Human TPO — rhTPO im, 300U/kg per day for 2 weeks, if response (Plt 30-100×100^g/L), taper to 300U/kg for twice per week until 6 weeks after delivery; if not response, drug withdrawal.
  Other Names: rhTPO
  Arms: Prednisone plus rhTPO

SUMMARY:
Randomized, open-label study to compare the efficacy and safety of prednisone plus recombinant human thrombopoietin (rhTPO) compared to prednisone monotherapy for the treatment of immune thrombocytopenia in pregnancy

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, randomized controlled trial of adults with ITP in pregnancy in China. Patients were randomized to prednisone plus rhTPO and prednisone monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-49;
2. Gestational weeks ≥20 weeks;
3. Platelet count <30×10^9/L, accompanied with or without bleeding symptoms;
4. Confirmed diagnosed, treatment-naive ITP in pregnancy;
5. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Secondary ITP such as drug-related thrombocytopenia;
2. Thrombocytopenia caused by viral infection (HIV, hepatitis B or hepatitis C); Other autoimmune diseases (including positive anti-nuclear antibodies, positive anti-cardiolipin antibodies, positive lupus anticoagulant factors, and positive Coombs) with severe heart, kidney, liver or respiratory dysfunction;
3. Severe immunodeficiency;
4. Myelodysplastic or myeloid fibrosis;
5. History of malignancy.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Response | day 14
  Response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Platelet counts at delivery | At delivery
  Platelet counts at delivery

SECONDARY OUTCOMES:
Number of patients with bleeding | During treatment（up to 6 weeks after delivery）
  Number of patients with bleeding symptome
Number of patients with adverse events | During treatment（up to 6 weeks after delivery）
  Number of patients with adverse events
Platelet counts of newborns | at delivery
  Platelet counts of newborns
Number of newborns with adverse events | During treatment（up to 6 weeks after delivery）
  Number of newborns with adverse events
Loss of response | During treatment（up to 6 weeks after delivery）
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-hui Zhang, Professor, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, China